CLINICAL TRIAL: NCT06074523
Title: Psychometric Testing: Cued vs. Learned Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9R15EY030247-01A1 (NIH)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: attention
MeSH Terms: interventions — Self Report

STUDY DESIGN:
Intervention Model Description: Within-subjects measures, correlational analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Attention and Working Memory Tests (Experimental): All participants will complete a series of behavioral tasks, including cued visual search with positive (target color), negative (distractor color) and neutral (baseline) cues, learned visual search with a repeated salient distractor color, a visual working memory capacity task, and a daily life inattentive traits questionnaire (self-report). Single Arm.
  Interventions: Behavioral: Behavioral Measurement and self-report

INTERVENTIONS:
Behavioral: Behavioral Measurement and self-report — Measurements of behavioral performance and self-report

SUMMARY:
In this line of research, the researchers are examining whether performance on a cued attentional suppression (ignoring) task is related to performance on a learned attentional suppression task. In addition, these measures are related to the capacity of working memory and every day inattentive traits.

DETAILED DESCRIPTION:
This is a behavioral study. The researchers will measures performance on multiple tasks. 1) a cued attentional suppression task, where participants are told the color of the item they are supposed to ignore on each trial. 2) a learned attentional suppression task, where participants learn over experience that a particular color is not the target. 3) a visual working memory capacity measurement 4) an inattentive trait report task, where participants report their experiences of inattention during their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected-to-normal visual acuity, normal color vision

Exclusion Criteria:

* age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Carlisle, PhD, Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymous behavioral performance data will be available for other researchers upon request
Supporting Information: Study Protocol, Analytic Code
Time Frame: Upon publication of the work, for at least 5 years
Access Criteria: Request

REFERENCES:
- [Background] Arita JT, Carlisle NB, Woodman GF. Templates for rejection: configuring attention to ignore task-irrelevant features. J Exp Psychol Hum Percept Perform. 2012 Jun;38(3):580-4. doi: 10.1037/a0027885. Epub 2012 Apr 2. PMID 22468723

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Attention and Working Memory Tests
Started | 75
Completed | 65
Not Completed | 10
Not completed — missing data in one condition, participant failed to fill out all data forms | 9
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Attention and Working Memory Tests
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.1 (1.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 56
  More than one race | 3
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Button Press Reaction Time
Description: Reaction times on visual search task with positive, negative, and neutral cues
Time Frame: 1 day
Population: 21 participants were excluded for either bad accuracy in one of the cognitive tasks (n = 11) or for incomplete data recording (n = 10).
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Attention and Working Memory Tests
Number analyzed (Participants) | 54
Seconds
  Neutral Condition | 1.86 (.77)
  Negative Condition | 1.53 (.57)
  Positive Condition | 1.29 (.49)
Statistical Analysis 1: Comparison: Attention and Working Memory Tests; Comparing Cued Suppression Task; Positive, Negative, and Neutral Cue condtions; Test type: Equivalence — Comparing three conditions in a basic science experiment in healthy adults; p < .001, ANOVA; partial eta squared = .81

2. Primary Outcome: Learned Suppression Task
Description: Reaction times on visual search task no salient distractor and learned salient distractor
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Reaction time (seconds)
Arm/Group | Attention and Working Memory Tests
Number analyzed (Participants) | 54
Reaction time (seconds)
  Singleton Absent condition | 1.014 (.315)
  Singleton Present condition | 1.001 (.294)
Statistical Analysis 1: Comparison: Attention and Working Memory Tests; Comparing performance on target absent and target present trials; Test type: Equivalence — P<.05 criterion; p = .08, t-test, 2 sided; cohen's d = .24

3. Primary Outcome: Visual Working Memory Capacity
Description: Visual Working Memory Capacity- Change Localization; Estimate of number of items maintained in working memory
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of items remembered
Arm/Group | Attention and Working Memory Tests
Number analyzed (Participants) | 54
Number of items remembered | 2.85 (.70)
Statistical Analysis 1: Comparison: Attention and Working Memory Tests; Relationship between Cued Attention Negative Cue Benefit (Neutral Cue RT- Negative Cue RT) and working memory capacity; Test type: Other; p = .007, correlation; Slope = -.37, 95% CI 2-sided [-0.5803 to -0.1135]

4. Primary Outcome: Inattentive Traits Subscale of Adult Attention Deficit Hyperactivity Disorder (ADHD) Self Report Scale
Description: Adult Attention Deficit Hyperactivity Disorder (ADHD) Self Report Scale (used on healthy adults), Inattentive Traits subscale. Higher values indicate more ADHD-like inattentive trait symptoms (0-45).
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Attention and Working Memory Tests
Number analyzed (Participants) | 54
units on scale | 18.1 (5.40)
Statistical Analysis 1: Comparison: Attention and Working Memory Tests; Correlation of Inattentive Traits subscale and learned suppression (difference in RT between target absent and target present trials); Test type: Other; p = .046, correlation; Slope = -.27, 95% CI 2-sided [-0.5015 to -0.002414]

ADVERSE EVENTS:
Time Frame: Participants were monitored during the testing session, which occurred during one day.
Arm/Group | Attention and Working Memory Tests
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 1/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attention and Working Memory Tests (N=75)
Participant Migraine (Nervous system disorders) | 1 (1) — Participant reported a migraine during the testing session, and chose to withdraw.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT06074523/Prot_SAP_ICF_000.pdf